CLINICAL TRIAL: NCT05328258
Title: A Phase 3 Randomised Double-Blinded Placebo-Controlled Study of Use of GnRHa During Chemotherapy for Fertility Protection of Young Women and Teenagers With Cancer
Brief Title: Use of GnRHa During Chemotherapy for Fertility Protection
Acronym: ProFertil
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kenny Rodriguez-Wallberg (Other)
Responsible Party: Sponsor-Investigator, Kenny Rodriguez-Wallberg, Adjunct professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProFertil
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer Female; Acute Leukemia; Lymphoma; Osteosarcoma; Soft Tissue Sarcoma; Ewing Sarcoma
Keywords: Fertility protection of young women receiving chemotherapy
MeSH Terms: conditions — Lymphoma; Osteosarcoma; Sarcoma; Sarcoma, Ewing | interventions — Triptorelin Pamoate

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, double-blinded, placebo-controlled, phase 3 study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects are randomised to triptorelin (active arm) or placebo (control) given in parallel to the chemotherapy treatment for the cancer diagnosis. All personnel involved in the study, and subjects, except personnel preparing triptorelin/placebo at the local site and an unblinded monitor, will be blinded during the study. Unblinded research nurse at each site will prepare blinded triptorelin/placebo to subjects and a web-based randomisation system will be used to allocate of blinded triptorelin/placebo to subjects at randomisation and drug dispense during the treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Triptorelin (Experimental): Triptorelin given intramuscularly once every month or every third month during gonadotoxic chemotherapy treatment.
  The dose is ether 11.25 mg triptorelin given for subjects having at least 3 months gonadotoxic treatment, OR 3.75 mg for subjects during one-month of gonadotoxic treatment
  Interventions: Drug: Triptorelin Embonate
- Arm B: Placebo (Placebo Comparator): Placebo, 0.9% sodium chloride, given intramuscularly once every month or every third month during gonadotoxic chemotherapy treatment.
  The dose will be provided both as one injection compensating for 3 months' effect and one injection compensating for 1 month' effect to maintain the study blind.
  Interventions: Drug: Sodium Chloride solution 0.9%

INTERVENTIONS:
Drug: Triptorelin Embonate — 11.25 mg will be given for subjects having at least 3 months gonadotoxic treatment, one injection of 11.25 mg will compensate for 3 months' effect of the study drug.
  3.75 mg will be given for subjects during one-month of gonadotoxic treatment, one injection of 3.75 mg will compensate for 1 month' effect of the study drug.
  Other Names: Pamorelin
  Arms: Arm A: Triptorelin
Drug: Sodium Chloride solution 0.9% — One injection compensating for 3 months' effect OR one injection compensating for 1 month' effect to maintain the study blind.
  Other Names: Placebo
  Arms: Arm B: Placebo

SUMMARY:
Many cytotoxic drugs may harm the fertility of young women treated for cancer. The aim of the study is to investigate if the Gonadotropin-Releasing Hormone agonist (GnRHa) during cancer treatment can preserve the fertility of young female cancer subjects.

Approximately 300 women with newly diagnosed breast cancer and up to 200 women with newly diagnosed lymphoma, acute leukemias or sarcomas will be recruited before start of cancer treatment.

The patients will be randomised in between treatment with triptorelin (experimental) or placebo (control) intramuscularly a 1:1 ratio during chemotherapy. The injections may be given once monthly or once three months depending on type of chemotherapy given. Randomisation and study drug is blinded, neither investigator, research nurse nor patient will know if it is active drug or placebo. The only person who knows is the nurse preparing the injection.

Patients will be followed up to 5 years after end of treatment with physical examinations, vital signs, biochemical markers, bone mineral density exams, ultrasound for antral follicle counts and ovarian doppler flow, concomitant medications, adverse events and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Breast cancer or acute leukemias, lymphomas (Hodgkin and non-Hodgkin) or sarcomas (osteo, soft tissue and Ewing) confirmed by histology and assigned for diseace-specific chemotheraphy
* Confirmed menarche
* ECOG performance status 0-1
* Adequate bone marrow, renal, hepatic and cardiac functions and absence of other uncontrolled medical or psychiatric disorders

Exclusion Criteria:

* Demonstrated premature ovarian failure at time of randomization according to clinical or biochemical data
* Previous or planned bilateral oophorectomy
* Pregnancy or breastfeeding at time of start of chemotherapy
* Other malignancy diagnosed within the last five years
* Uncontrolled hypertension, heart, liver, kidney related or other uncontrolled medical or psychiatric disorders including previous or current diagnosis of anorexia
* Known osteoporosis
* Known low platelet count with increased bleeding risk or refractory thrombocytopenia in subjects with acute leukemias
* Known or suspected allergy against triptorelin
* Direct radiation of the gonads previous or planned (TBI allowed)
* Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation

Ages: 14 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Müllerian Hormone (AMH) levels in women with breast cancer | 12 months after end of gonadotoxic chemotherapy and study drug treatment
  To estimate the changes in ovarian reserve following chemotherapy for treatment of cancer with or without GnRHa by determination of the AMH relative to AMH levels at EoT in women with breast cancer.

SECONDARY OUTCOMES:
Anti-Müllerian Hormone (AMH) levels in women with acute leukemias, lymphomas and sarcomas. | 12 months after end of gonadotoxic chemotherapy and study drug treatment
  To estimate the changes in ovarian reserve following chemotherapy for treatment of cancer with or without GnRHa by determination of the AMH relative to AMH levels at EoT in women with acute leukemias, lymphomas and sarcomas.
Changes in ovarian reserve with or without Gonadotropin-Releasing Hormone agonist (GnRHa) by determination of the antral follicle counts (AFC) | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months) and at 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT
  Changes in AFC in women with breast cancer and with acute leukemia, lymphoma and sarcoma respectively
Changes in ovarian reserve with or without GnRHa by longitudinal observation of AMH levels | At 6 months, 2 years, 3 years, 4 years and 5 years after EoT.
  The difference in recovery of AMH levels between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively
The proportion of females with or without GnRHa that develop ovarian insufficiency by determination of follicle stimulating hormone (FSH), inhibin and estradiol | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of FSH, inhibin and estradiol between the GnRHa group and the placebo group
Impact of body mass index (BMI) (Kg/m2) on changes in ovarian reserve with or without GnRHa | At Baseline, during treatment, at end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  longitudinal observation of AMH levels, FSH, inhibin and estradiol
Impact of use of contraceptives (yes/no) in changes of ovarian reserve with or without GnRHa | At Baseline, during treatment visits (every 1-3 months of gonadotoxic treatment), at end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  longitudinal observation of AMH levels, FSH, inhibin and estradiol
Impact of endocrine adjuvant therapy (yes/no) in changes of ovarian reserve with or without GnRHa | At Baseline, during treatment visits (every 1-3 months of gonadotoxic treatment), at end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  longitudinal observation of AMH levels, FSH, inhibin and estradiol
The effect of GnRHa with or without GnRHa on ovarian blood supply | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of blood flow to the ovarian artery (right and left Doppler flow) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively
The proportion of females with or without GnRHa that develop amenorrhea (no menstruations) | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of the proportion that develop amenorrhea (no menstruations) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively
Pregnacy wish after cancer treatment in women with or without GnRHa who attempt pregnancy during follow-up | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of of pregnancy wish (Study specific questionaire) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Fertility and childbirth after cancer treatment in women with or without GnRHa who attempt pregnancy during follow-up | At end of chemotherapy (corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of pregnancy attempts (Study specific questionaire) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Fertility and childbirth after cancer treatment in women with or without GnRHa who attempt pregnancy during follow-up | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of pregnancy outcome between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Health-related quality of life (EORTC QLQ C30) | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of validated outcome on health-related QoL (EORTC QLQ C30) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Health-related quality of life (FSFI) | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of validated outcome of sexuality and reproductive health (Female Sexual Function Index (FSFI)) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Health-related quality of life (HAD) | At end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months), and 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Comparison of validated outcome on health-related QoL (Hospital Anxiety and Depression Scale (HAD)) between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
The development of co-morbidities during follow-up and bone mineral density | At baseline, at end of gonadotoxic chemotherapy (EoT; corresponding to Baseline+2-11 months) and 12 months and 5 years after EoT
  Comparison of bone mineral density between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Disease-specific oncologic outcomes: disease-free survival | At 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Investigation of disease-free survival between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Disease-specific oncologic outcomes: Recurrence rate | At 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Investigation of recurrence rate between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.
Disease-specific oncologic outcomes: overall survival | At 12 months, 2 years, 3 years, 4 years and 5 years after EoT.
  Investigation of overall survival between the GnRHa group and the placebo group in women with breast cancer and in women with acute leukemia, lymphoma and sarcoma respectively.

CONTACTS AND LOCATIONS:
Locations (17):
- Sweden (17):
  - Center for Pediatric Cancer, Queen Silvia Hospital for Children and Youth, Gothenburg
  - Center for Pediatric Oncology, Akademiska Hospital, Gothenburg
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Department of Hematology, Skåne University Hospital, Lund
  - Department of Oncology, Skåne University Hospital, Lund
  - Department of Pediatric Oncology, Skåne University Hospital, Lund
  - Department of Oncology, Örebro University Hospital, Örebro
  - Karolinska Univeristy Hospital, Breast Centre, Stockholm
  - Department of Hematology and coagulation, Sahlgrenska University Hospital, Stockholm
  - Department of Hematology, Capio ST. Göran Hospital, Stockholm
  - Department of Internal Medicine, Södersjukhuset, Stockholm
  - Department of Oncology, Capio ST. Göran Hospital, Stockholm
  - Department of Oncology, Södersjukhuset, Stockholm
  - Division of Hematology, Department of Medicine Huddinge, Karolinska Institutet, Stockholm
  - Karolinska University Hospital, Hematology, Stockholm
  - Karolinska University Hospital, High Specialised Pediatric Medicine, Stockholm
  - Department of Oncology, Norrlands University Hospital, Umeå

IPD SHARING:
Plan to Share IPD: No
The identity of the individual participants is protected by GDPR through the The Swedish Authority for Privacy Protection as regulated by the informed consent and any data sharing must be in accordance with their regulations. We can thus only share IPD that underlie the results reported in this study (text, tables, figures, and appendices), after full anonymization of the data.
  After completion of the study the protocol, informed consent form and statistical analysis plan will be available.
  Requests for additional analyses or to access the anonymized datasets should be directed to kenny.rodriguez-wallberg@ki.se. Information will be available upon reasonable request to the sponsor and if in correspondence with the proposed research in the signed informed consent e.g to achieve aims in the approved proposal.

REFERENCES:
- [Derived] Rodriguez-Wallberg KA, Nilsson HP, Bergh J, Malmros J, Ljungman P, Foukakis T, Stragliotto CL, Friman EI, Linderholm B, Valachis A, Andersson A, Harrysson S, Vennstrom L, Frisk P, Morse H, Eloranta S. ProFertil study protocol for the investigation of gonadotropin-releasing hormone agonists (GnRHa) during chemotherapy aiming at fertility protection of young women and teenagers with cancer in Sweden-a phase III randomised double-blinded placebo-controlled study. BMJ Open. 2023 Dec 9;13(12):e078023. doi: 10.1136/bmjopen-2023-078023. PMID 38070906